CLINICAL TRIAL: NCT06392659
Title: A Phase 1, Open-label Study Evaluating the Effect of VX-993 on the Pharmacokinetics of Midazolam, and the Effect of Itraconazole and Gemfibrozil on the Pharmacokinetics of VX-993, in Healthy Adults
Brief Title: A Phase 1, Open-label Study Evaluating the Pharmacokinetics and Drug-drug Interaction of VX-993 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX24-993-004
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Gemfibrozil; Itraconazole; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Midazolam (Experimental): Participants will receive a single dose of Midazolam in absence and presence of VX-993.
  Interventions: Drug: VX-993; Drug: Midazolam
- Part B: Itraconazole (Experimental): Participants will receive a single dose of VX-993 on Day 1 and Itraconazole once daily (qd) on Days 7 through Day 15. On Day 10 participants will receive Itraconazole followed by VX-993.
  Interventions: Drug: VX-993; Drug: Itraconazole
- Part C: Gemfibrozil (Experimental): Participants will receive a single dose of VX-993 on Day 1 and Gemfibrozil every 12 hours (q12d) on Days 7 through Day 15. On Day 10 participants will receive Gemfibrozil followed by VX-993.
  Interventions: Drug: VX-993; Drug: Gemfibrozil

INTERVENTIONS:
Drug: VX-993 — Suspension for Oral Administration.
Drug: Gemfibrozil — Tablets for Oral Administration.
  Arms: Part C: Gemfibrozil
Drug: Itraconazole — Capsules for Oral Administration.
  Arms: Part B: Itraconazole
Drug: Midazolam — Solution for Oral Administration.
  Arms: Part A: Midazolam

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), drug-drug interaction, and safety and tolerability of VX-993 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg
* Nonsmoker or ex-smoker for at least 3 months before the first study drug dose

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug.
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of Midazolam in Absence or Presence of VX-993 | Pre-dose up to Day 15
Part A: Maximum Observed Plasma Concentration (Cmax) of 1-Hydroxy-Midazolam in Absence or Presence of VX-993 | Pre-dose up to Day 15
Part A: Area Under the Concentration Versus Time Curve (AUC) of Midazolam in Absence and Presence of VX-993 | Pre-dose up to Day 15
Part A: Area Under the Concentration Versus Time Curve (AUC) of 1-Hydroxy-Midazolam in Absence and Presence of VX-993 | Pre-dose up to Day 15
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-993 in Absence or Presence of Itraconazole | Pre-dose up to Day 27
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-993 in Absence or Presence of Itraconazole | Pre-dose up to Day 27
Part C: Maximum Observed Plasma Concentration (Cmax) of VX-993 in Absence or Presence of Gemfibrozil | Pre-dose up to Day 27
Part C: Area Under the Concentration Versus Time Curve (AUC) of VX-993 in Absence or Presence of Gemfibrozil | Pre-dose up to Day 27

SECONDARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 30
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 27
Part C: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 27

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing